CLINICAL TRIAL: NCT02736539
Title: Clinical Trial of CBS-2004 in Prevention of Travelers' Diarrhea
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Commercial strategy
Sponsor: Clasado Biosciences Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IDCRP-080
Record Dates: First submitted 2016-04-05; First posted 2016-04-13 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Traveler's Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): galacto-oligosaccharides
  Interventions: Drug: CBS 2004 (galacto-oligosaccharides)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBS 2004 (galacto-oligosaccharides) — CBS 2004 active treatment
  Arms: Active
Drug: Placebo — Placebo treatment
  Arms: Placebo

SUMMARY:
This study is designed as a randomized double-blinded treatment trial among travelers' to geographical areas with moderate-severe rates of traveler's diarrhea. Travelers will be randomized to receive CBS 2004 or masked placebo to be taken daily while traveling. The test article or placebo will be taken starting 7 days prior to travel.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, 18 years old or older
2. Travel on moderate-high risk itinerary for traveler's diarrhea for minimum of 14 days and maximum of 6 weeks travel
3. Able to comply with study and follow-up procedures
4. Subjects willing and able to enter data in the diary card
5. An IRB approved informed consent form is signed and dated
6. Subjects must have adequate general health (as determined by investigators)
7. Women: Non-nursing and negative urine/serum pregnancy test with understanding through informed consent process to avoid pregnancy during the study while on the study drug. Should an individual have a documented surgical sterilization in her medical record, a pregnancy test will not be required. If a volunteer becomes pregnant during the study, the Principal Investigator (PI) will notify the study research monitor and the Institutional Review Boards (IRBs). The pregnancy outcome will be followed per IRB and other regulatory requirements.

Exclusion Criteria:

1. Allergy to investigational product
2. History of functional bowel disorder (including IBS)
3. Chronic intestinal disease (ulcerative colitis, crohn's disease), post vagotomy diabetic autonomic neuropathy, malabsorption, short bowel syndrome, celiac disease, bacterial overgrowth due to blind loops, pancreatitis
4. Antibiotic use within 7 days prior to enrollment (except for malaria prophylaxis excluding doxycycline)
5. Use of other probiotics or prebiotics (outside of the study product) in the prior 3-weeks or intent to use during the study period. This includes the over-the-counter preparations of probiotics, prebiotics (including inulin, lactulose) or consumption of a bio-yogurt product.
6. Lactose intolerant (allergies to dairy products).
7. Medications usage as deemed by the PI to interfere with GI function
8. Diarrheal illness within 7 days prior to enrollment
9. Subject has a concomitant disease or condition that could interfere with or for which treatment could interfere with the conduct of the study, or could in the opinion of the investigator increase the risk of adverse events (AEs) during the subject's participation in the study.
10. Use of any investigational or non-registered drug other than the study drug within 30 days preceding the study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-15 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Assess safety and tolerance by evaluating the adverse events reported with study drug and placebo during the period of prophylaxis and through the last clinic visit. | 7 weeks
To assess the effectiveness of CBS 2004 by evaluating the development of traveler's diarrhea (TD) with CBS-2004 versus placebo based on time to first unformed stool associated with a TD episode | 7 weeks

SECONDARY OUTCOMES:
Assess the number of work days lost due to diarrhea | 7 weeks
Assess percentages of subjects requiring treatment for diarrhea | 7 weeks
Assess total number of diarrheal days | 7 weeks

IPD SHARING:
Plan to Share IPD: Undecided